CLINICAL TRIAL: NCT06766916
Title: Crisugabalin Versus Pregabalin for Radiotherapy-Related Neuropathic Pain in Head and Neck Cancers: A Multicenter, Randomized, Open-Label, Non-Inferiority Trial
Brief Title: Crisugabalin for Radiotherapy-Related Neuropathic Pain
Acronym: CRYSTAL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-1020-02
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-02

CONDITIONS: Neuropathic Pain
Keywords: Head and Neck Cancers; Radiotherapy-Related Neuropathic Pain; Crisugabalin
MeSH Terms: conditions — Neuralgia; Head and Neck Neoplasms | interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Crisugabalin (Experimental): The initial dose is one Crisugabalin capsule (20 mg) taken twice daily. The dose will be gradually increased to the maximum tolerated dose or the maximum daily dose of three capsules (60 mg) taken twice daily.
  Interventions: Drug: Crisugabalin
- Pregabalin (Active Comparator): The initial dose is one capsule of Pregabalin (75 mg) taken twice daily. The dose will be gradually increased to the maximum tolerated dose or the maximum daily dose of four capsules (300 mg) taken twice daily.
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Crisugabalin — Days 1-14: Crisugabalin 40 mg/day, 20 mg twice daily, orally. Days 15-21: Increase dose to 80 mg/day, 40 mg twice daily. If not tolerated, maintain previous dose until the end of the treatment period.
  Days 22-28: Increase dose to 120 mg/day, 60 mg twice daily. If not tolerated, maintain previous dose until the end of the treatment period.
  Arms: Crisugabalin
Drug: Pregabalin — Days 1-7: Pregabalin 150 mg/day, 75 mg twice daily, orally. Days 8-14: Increase dose to 300 mg/day, 150 mg twice daily. Days 15-21: Increase dose to 450 mg/day, 225 mg twice daily. If not tolerated, maintain previous dose until the end of the treatment period.
  Days 22-28: Increase dose to 600 mg/day, 300 mg twice daily. If not tolerated, maintain previous dose until the end of the treatment period.
  Arms: Pregabalin

SUMMARY:
The purpose of this study is to evaluate whether Crisugabalin has similar efficacy compared to Pregabalin in reducing radiotherapy-related neuropathic pain (RRNP) in patients with head and neck cancers.

DETAILED DESCRIPTION:
The primary objective of this study is to determine whether Crisugabalin provides non-inferior pain relief compared to Pregabalin in patients with head and neck cancer experiencing radiotherapy-related neuropathic pain. The trial adopts a multicenter, randomized, open-label design, and the primary endpoint is the change in Numeric Rating Scale (NRS) pain scores from baseline to 4 weeks. The study aims to provide new evidence to support treatment strategies for this condition, which significantly affects patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily sign a written informed consent form.
2. Male or female patients aged ≥18 years with an expected survival of at least 5 months.
3. Histologically confirmed head and neck tumors treated with radiotherapy at least 6 months prior to screening.
4. Average NRS pain score ≥4 over 7 days during the screening period, with pain localized to nerve-innervated areas corresponding to the radiotherapy site, such as the head, face, neck, and arms.
5. Diagnosis of neuropathic pain persisting for at least 4 weeks, confirmed by two trained neurologists based on clinical history, symptoms, signs, and a Leeds Assessment of Neuropathic Symptoms and Signs (LANSS) score ≥12 (Chinese version).
6. Adequate cognitive and language abilities to communicate and complete study questionnaires.

Exclusion Criteria:

1. Severe abnormalities in hematological, hepatic, or renal function, as evidenced by:

   * Hematology: Neutrophil count <1.5×10⁹/L, platelet count <90×10⁹/L, or hemoglobin <100 g/L.
   * Liver function: Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3× upper limit of normal (ULN), or total bilirubin (TBIL) >1.5× ULN.
   * Renal function: Estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m² or undergoing dialysis.
   * Creatine kinase >2× ULN.
2. Chronic systemic diseases that may interfere with study participation, including but not limited to:

   * Severe cardiopulmonary diseases such as unstable angina, myocardial infarction, severe arrhythmia, WHO functional classification III-IV heart failure, uncontrolled hypertension (systolic BP >160 mmHg or diastolic BP >100 mmHg), or recurrent asthma.
   * Chronic gastrointestinal diseases, such as liver fibrosis, recurrent indigestion or diarrhea, or peptic ulcers.
   * Neurological or psychiatric conditions affecting pain assessment, including epilepsy, recurrent dizziness, headache, memory, or cognitive disorders; cerebrovascular accidents or transient ischemic attacks within 6 months of screening.
3. Known allergy to study drugs or chemically related compounds.
4. Current diagnosis of tumor recurrence or metastasis associated with tumor-related pain.
5. Neuropathic pain not caused by radiotherapy, such as postherpetic neuralgia, diabetic neuropathy, HIV-related neuropathy, spinal cord injury, or other neurological diseases.
6. Use of pregabalin/crisugabalin within 4 weeks before screening.
7. Pregnant, planning to become pregnant during the study, or breastfeeding. Participants and their partners unwilling to use reliable contraception (e.g., condoms, spermicides, intrauterine devices) from the time of consent until 28 days after the last dose of study medication.
8. Participation in any other clinical trial within 30 days prior to screening.
9. Any other condition deemed unsuitable for study participation by the investigator.
10. Use of prohibited medications within at least 5 half-lives of the drug before screening, with prohibition maintained throughout the study.
11. Previous use of pregabalin ≥300 mg/day or gabapentin ≥1200 mg/day deemed ineffective.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Rating Scale (NRS) Change | 4 weeks
  The change in NRS score from baseline to Week 4 of treatment. The NRS measures pain intensity on a scale of 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain.

SECONDARY OUTCOMES:
Numeric Rating Scale (NRS) Change | 1 week
  The change in NRS score from baseline to Week 1 of treatment. The NRS measures pain intensity on a scale of 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain.
Visual Analogue Scale (VAS) Change | 4 weeks
  The VAS measures pain intensity on a 0-100 mm scale, with 0 representing no pain and 100 representing the worst imaginable pain.
Hamilton Anxiety Scale (HAMA) and Hamilton Depression Scale (HAMD) scores | 4 weeks
  The HAMA and HAMD are used to evaluate anxiety and depressive symptoms, respectively.
Daily Sleep Interference Scale (DSIS) | 4 weeks
  The DSIS measures the impact of pain on sleep quality. Scores range from 0 (no interference) to 10 (complete interference).
Health Status According to EuroQol-5-Domain-5-Level health questionnaire (EQ-5D-5L) | 4 weeks
  The EQ-5D-5L assessed quality of life based on 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The participant was asked to 'check the ONE box that best describes your health TODAY,' choosing from 5 options (no problems, slight problems, moderate problems, severe problems, extreme problems) provided under each dimension.
  The health state index value is a single value on a scale from 0 to 100 scores indicating better health: 0 = indicating worst health and 100 = best imaginable health.
Response Rates | 4 weeks
  The proportion of patients achieving ≥30% and ≥50% reductions in NRS score from baseline to Week 4.
Short-Form McGill Pain Questionnaire (SF-MPQ) | 4 weeks
  Participants rate their pain in three parts of the questionnaire, which are combined into a single pain intensity score:
  Part 1 - fifteen descriptors of pain intensity, on a scale of 0 (none) to 3 (severe); Part 2 - the VAS, in which the participant rates pain on a 100 mm-long horizontal line, where 0 mm = no pain and 100 mm = worst possible pain; Part 3 - a present pain intensity index in which the participant rates present pain intensity on a scale of 0 (no pain) to 5 (most intense pain).
Patient Global Impression of Change (PGIC) | 4 weeks
  PGIC is a 7 point scale depicting a patient's rating of overall improvement, with 1 representing very much improved and 7 representing very much worse.

CONTACTS AND LOCATIONS:
Overall Officials: Yamei Tang, M.D., PhD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (11):
- China (11):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affillated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - The Affiliated Brain Hospital, Guangzhou Medical University, Guangzhou, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Cancer Hospital (Affiliated Cancer Hospital of ZhengzhouUniversity), Zhengzhou, Henan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan Brain Hospital, Changsha, Hunan
  - Changsha Central Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available from Principal Investigator upon reasonable request 6 months after the trial completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after the trial completion
Access Criteria: The IPD will be available from Principal Investigator upon reasonable request.